CLINICAL TRIAL: NCT02550275
Title: Social Cognition in Huntington's Disease: Cognitive Study and Functional and Morphological Imaging
Acronym: COSIMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOI 201409
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2015-09

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Neuropsychological Tests

ARMS (3):
- presymptomatic patient (Other): patient with Unified Huntington's Disease Rating Scale (UHDRS) < 5
  Interventions: Behavioral: neuropsychological test; Radiation: MRI
- symptomatic patient (Other): patient with Unified Huntington's Disease Rating Scale (UHDRS) > 5
  Interventions: Behavioral: neuropsychological test; Radiation: MRI
- controls (Other): unaffected patient with Huntington's disease
  Interventions: Behavioral: neuropsychological test; Radiation: MRI

INTERVENTIONS:
Behavioral: neuropsychological test
Radiation: MRI

SUMMARY:
Huntington's disease is a rare genetic neurodegenerative disease. It is accompanied by movement disorders, cognitive and behavioral. The social behavior of patients are changed, affecting interpersonal relationships. Patients with Huntington's disease are described as self-centered, lacking sympathy and empathy and mentally inflexible. These behavioral problems can be a major source of anxiety for patients and their families. These disorders also have a negative impact cognitive and motor symptoms as well as the functional abilities and the quality of life of patients and their entourage. Authors have suggested that these problems could be related inter alia to social cognition disorders. This concept refers to a set of skills and emotional and social experiences that regulate relations between individuals and can explain the behavior of individuals and groups. The objective is to evaluate disorders of social cognition, which may account for behavioral changes in Huntington's disease.

ELIGIBILITY:
Inclusion Criteria:

For all particpipants

* Patient gave its written consent
* between 20 and 70 years
* School level : at least 7 years
* native language: french

For presymptomatic patient

* Huntington's disease diagnosed with abnormal number of CAG repeats: 36 < nucleotide expansion (CAG)
* Unified Huntington Disease Rating Scale moteur ≤ 5

For symptomatic patient

* Huntington's disease diagnosed with abnormal number of CAG repeats: 36 < nucleotide expansion (CAG)
* Unified Huntington Disease Rating Scale moteur > 5

Exclusion Criteria:

* No national health insurance affiliation
* Being under guardianship
* Meeting brain MRI exclusion criteria (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body, Renal failure, hypersensitivity of Gadolinium) or refusing MRI
* Pregnant or lactating women
* Patient with involuntary movement hampering the realization of MRI

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
the achievement of social cognition process in Huntington's disease using the total score of the scale 15-TOM | 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: SCHERER GAGOU, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France